CLINICAL TRIAL: NCT05291949
Title: Comparison of Intraoperative Heart Rate and Respiratory Rate Acquired Via ATLASense Raphael Polymonitor and Standard Intraoperative Monitors
Brief Title: Comparison of Intraoperative HR and RR Acquired Via ATLASense Raphael PolyMonitor and Standard Intraoperative Monitors
Acronym: ATLASense
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Trevor J. Szymanski MD, MBA, Senior Staff Anesthesiologist, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14139
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Results first posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Intraoperative Monitoring
Keywords: heart rate; respiratory rate; blood pressure; temperature

STUDY DESIGN:
Intervention Model Description: Each patient receives monitoring by all standard intraoperative monitors in addition to monitoring by the ATLASense RAPHAEL PolyMonitor during their surgery.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- ATLASense RAPHAEL monitoring (Experimental): All patients receive monitoring by ATLASense RAPHAEL PolyMonitor for duration of surgery.
  Interventions: Device: ATLASense RAPHAEL PolyMonitor

INTERVENTIONS:
Device: ATLASense RAPHAEL PolyMonitor — All patients will be monitored using the ATLASense RAPHAEL PolyMonitor during their surgery.

SUMMARY:
The aim of this observational comparison study is to compare the HR and respiratory RR of intraoperative surgical patients simultaneously recorded by standard intraoperative monitors and the ATLASense RAPHAEL PolyMonitor. A second aim is to determine the extent of data loss and data gap duration, and validate the PolyMonitor alert system for tachycardia and bradycardia. Additional parameters of non-invasive blood pressure (NIBP) and body temperature will also be compared between the PolyMonitor and standard intraoperative monitors. Finally, this study will provide insight into the logistics of intraoperative use of the PolyMonitor.

DETAILED DESCRIPTION:
The ATLASense Raphael PolyMonitor will be placed on the patient's left chest mid sternal line in the operating room. Traditional physiologic monitors described above will also be placed on the patient in the operating room. Data will be collected via the ATLASense system and through the traditional operating room monitors, and this data will be time matched through synchronization of the monitors post hoc. The time matched data pairs will undergo statistical analysis post hoc. It is anticipated that this study will validate the intraoperative HR and RR measured through the ATLASense Raphael PolyMonitor, providing adequate data points for statistical analysis with 95% limits of agreement, bias, and data loss/gaps. Success is also the logistical lessons learned for using this monitor in the intraoperative setting.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Adult males or females (above the age of 18)
* Scheduled to undergo general anesthesia during elective surgery

Exclusion Criteria:

* Pregnant adult female
* Thoracic surgery
* Left lateral decubitus positioning required during procedure
* Surgery involving the left flank, or requiring surgical field involving the left flank
* Surgery involving the left chest, or requiring surgical field involving the left chest
* Allergy to adhesives
* Open wound, rash, or sore involving the left chest
* Presence of cardiac defibrillator, or pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Szymanski, MD, MBA, Principal Investigator — Medical Co-Director, Surgical Services, Division Head, Cardiac Anesthesia
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ATLASense RAPHAEL Monitoring
Started | 70
Completed | 66
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | ATLASense RAPHAEL Monitoring
Number analyzed (Participants) | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 52
  >=65 years | 18
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 60 [46 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 48
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 70

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate (HR)
Description: Minute-by-minute heart rate measures taken by both the ATLASense RAPHAEL PolyMonitor and the standard intraoperative monitor
Time Frame: Entire duration of surgery
Population: This only includes participants who were enrolled after the interim analysis, and who had HR data available from the standard intraoperative monitors.
Measure: Mean (Standard Deviation); unit: Spearman Correlation Coefficient
Arm/Group | ATLASense RAPHAEL Monitoring
Number analyzed (Participants) | 42
Spearman Correlation Coefficient | 0.922 (0.074)
Statistical Analysis 1: Comparison: ATLASense RAPHAEL Monitoring; Test type: Other — Bland-Altman; Bland-Altman; Bias = 0.3; Lower 95% Limit of agreement (LoA) value = -0.34 Upper 95% LoA = 0.94

2. Primary Outcome: Respiratory Rate (RR)
Description: Minute-by-minute respiratory rate measures taken by both the ATLASense RAPHAEL PolyMonitor and the standard intraoperative monitor
Time Frame: Entire duration of surgery
Population: Only participants who were enrolled after the interim analysis was performed and who had respiratory rate data available from standard intraoperative monitors. (Note: Intraoperative data from standard monitors was unretrievable from EPIC for two of the subjects)
Measure: Mean (Standard Deviation); unit: Weighted Spearman Correlation Coefficien
Arm/Group | ATLASense RAPHAEL Monitoring
Number analyzed (Participants) | 40
Weighted Spearman Correlation Coefficien | 0.714 (0.168)

3. Secondary Outcome: Gaps in Data Collection
Description: Length and frequency of gaps in data collection when the ATLASense RAPHAEL PolyMonitor or standard intraoperative monitors did not collect data.
Time Frame: Entire duration of surgery
Population: All participants who had HR or RR data available from standard intraoperative monitors.
Measure: Number; unit: percent of data loss
Arm/Group | ATLASense RAPHAEL Monitoring
Number analyzed (Participants) | 66
percent of data loss | 15.5

4. Secondary Outcome: Blood Pressure (Mean Arterial Pressure)
Description: Minute-by-minute blood pressure measures taken by both the ATLASense RAPHAEL PolyMonitor and the standard intraoperative monitor
Time Frame: Entire duration of surgery
Population: All patients who received continuous blood pressure monitoring via an arterial line for the duration of their procedure.
Measure: Mean (Standard Deviation); unit: Weighted Spearman Correlation Coefficien
Arm/Group | ATLASense RAPHAEL Monitoring
Number analyzed (Participants) | 14
Weighted Spearman Correlation Coefficien | 0.065 (0.113)

5. Secondary Outcome: Core Body Temperature
Description: Minute-by-minute core body temperature measures taken by both the ATLASense RAPHAEL PolyMonitor and the standard intraoperative monitor
Time Frame: Entire duration of surgery
Population: All patients enrolled after the interim analysis and who had temperature data available from standard intraoperative monitors. (Note: Intraoperative data from standard monitors was unretrievable from EPIC for two of the subjects)
Measure: Mean (Standard Deviation); unit: Weighted Spearman Correlation Coefficien
Arm/Group | ATLASense RAPHAEL Monitoring
Number analyzed (Participants) | 40
Weighted Spearman Correlation Coefficien | 0.158 (0.358)

ADVERSE EVENTS:
Time Frame: For the duration of procedure
Arm/Group | ATLASense RAPHAEL Monitoring
All-Cause Mortality (participants affected / at risk) | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT05291949/Prot_SAP_000.pdf